CLINICAL TRIAL: NCT05226741
Title: Design of Protective Headgear for Patients Who Have Undergone a Craniectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021/00540
Record Dates: First submitted 2022-01-13; First posted 2022-02-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Craniectomy
Keywords: helmet, protection,

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Head protection (Experimental): Participants are given a form of head protection
  Interventions: Device: Head protection device

INTERVENTIONS:
Device: Head protection device — The participants are fitted with a form of head protection over the craniectomy and provide feedback on design, use, and comfort

SUMMARY:
To design and create wearable head protection to be worn on a patient's head following a neurosurgical procedure (namely craniectomy and craniotomy

DETAILED DESCRIPTION:
After being given informed consent, all participants will undergo the fitting and trial of a specially designed head protection for 6 weeks. Week 1 participants will be assessed and clinical data obtained on participants condition with the head protection fitted during the same session. Participants will return after 3 weeks for review and adjustment and again at the 6 week interval where they will also be given a questionnaire to fill up regarding their use and comfort.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are eligible if they are 21 years or above and have had a DC >30 days, no wounds, able to understand simple commands and have a primary caregiver

Exclusion Criteria:

* Exclusion criteria are patients with severe cognitive impairment, wounds, > unilateral DC, no caregiver

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction Survey | 6 weeks after receiving their head protection fitting
  A survey to assess Satisfaction with device

SECONDARY OUTCOMES:
Euro Quality of Life - 5 Dimensions (EQ-5D) | 6 weeks after receiving their head protection fitting
  Quality of life survey. The higher the score from 0-5 for each dimension, the higher the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Trevor Binedell, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Anonymised Information will be published in a journal once completed

REFERENCES:
- [Background] Colasante C, Sanford Z, Castro N, Bartels MN. Custom Fabrication of a 3-Dimensionally Printed Helmet for Improved Socialization and Subjective Self-Assessment in a Case of Acquired Cranial Defect: A Case Presentation. PM R. 2018 Jun;10(6):671-674. doi: 10.1016/j.pmrj.2017.11.005. Epub 2017 Dec 30. PMID 29291381
- [Background] Lucano LRG, Brambila FJP, Perez JE, Rosales PH. Customized Low-Cost 3D Printed Helmet as a Temporary Measure for a Patient with Acrania. Indian J Plast Surg. 2019 May;52(2):252-253. doi: 10.1055/s-0039-1696077. Epub 2019 Sep 12. No abstract available. PMID 31602146